CLINICAL TRIAL: NCT06645288
Title: The Use of an Emergency Reflex Action Drill in Emergency Surgical Airway
Brief Title: The Evaluation of Training an Emergency Reflex Action Drill in the Emergency Surgical Airway in Dutch Paramedics
Acronym: ERAD-ESA
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Iscander M Maissan, Dr. I.M. Maissan MD PhD, Erasmus Medical Center
Other Study IDs: MEC-2024-0388
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Emergency Medical Services; Airway Management; Cricothyroidotomy; Prehospital; Prehospital Emergency Medical Services; Prehospital Setting; Self Confidence
Keywords: Emergency Reflex Action Drill; Emergency Surgical Airway; Emergency Medical Services; Prehospital; Cricothyrotomy; Coniotomy; Porcine model; 3D model; Self-confidence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Emergency Reflex Action Drill — Emergency Reflex Action Drill in performing Emergency Surgical Airway

SUMMARY:
The goal of this observational study is to learn about the effects of training an Emergency Reflex Action Drill (ERAD) for Emergency Surgical Airway (ESA) in Dutch paramedics. The main question it aims to answer is:

- Does training an ERAD improves self-confidence in performing an ESA in Dutch paramedics Participants will fill out a questionnaire directly before and after the training. To investigate long-term effects, they will be asked to fill out a questionnaire after 2 till 3 months and after one year.

ELIGIBILITY:
Inclusion Criteria:

* Registered Dutch paramedic
* Ambulance driver on Advanced Life Support Ambulance
* Participant in the two-day trauma course.

Exclusion Criteria:

* Medium care ambulance paramedic

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include Dutch paramedics attending a course. Dutch paramedics are all registered nurses with a background in Intensive Care, Anaesthesiology or Emergency Care. EMS training comprises an additional nine months of training and assessments, to be concluded with a final exam. Also, ambulance drivers of ambulances providing advanced life support (excluding medium care ambulances) who participate in the course are eligible to participate due to their supporting role in airway management.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Self-confidence | Baseline, pre-training up to immediately after the training
  Increase/decrease/no difference in self-confidence from baseline, assessed by a five-point Likert-scale of paramedics in performing an Emergency Surgical Airway

SECONDARY OUTCOMES:
Training model | Immediately after the training
  Difference in effect on self-confidence between two training models used during the ESA-ERAD training, assessed by a five-point Likert-scale.
Self-confidence real life cases | Through study completion, an average of 1 year
  Increase/decrease/no difference in self-confidence assessed by a five-point Likert-scale and correctly placed emergency surgical airway in real-life cases reported by paramedics at any time point after the ESA-ERAD training, up to an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Iscander M Maissan, Principal Investigator — Erasmus Medical Center
Locations (1):
- Academie van Ambulancezorg, Harderwijk, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning after 6 months after publication, ending 10 years after publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Unver V, Basak T, Watts P, Gaioso V, Moss J, Tastan S, Iyigun E, Tosun N. The reliability and validity of three questionnaires: The Student Satisfaction and Self-Confidence in Learning Scale, Simulation Design Scale, and Educational Practices Questionnaire. Contemp Nurse. 2017 Feb;53(1):60-74. doi: 10.1080/10376178.2017.1282319. Epub 2017 Feb 10. PMID 28084900
- [Background] Armstrong L, Harding F, Critchley J, McNarry AF, Myatra SN, Cooper R, Baker PA; World Airway Management Meeting 2015 Education Group. An international survey of airway management education in 61 countriesdagger. Br J Anaesth. 2020 Jul;125(1):e54-e60. doi: 10.1016/j.bja.2020.04.051. Epub 2020 May 20. PMID 32444066
- [Background] Iverson K, Riojas R, Sharon D, Hall AB. Objective comparison of animal training versus artificial simulation for initial cricothyroidotomy training. Am Surg. 2015 May;81(5):515-8. PMID 25975338
- [Background] Gustafson ML, Hensley B, Dotson M, Broce M, Tager A. Comparison of Manikin Versus Porcine Trachea Models When Teaching Emergent Cricothyroidotomy Among Emergency Medicine Residents. AEM Educ Train. 2019 Apr 7;3(3):280-285. doi: 10.1002/aet2.10333. eCollection 2019 Jul. PMID 31360821
- [Background] Cho J, Kang GH, Kim EC, Oh YM, Choi HJ, Im TH, Yang JH, Cho YS, Chung HS. Comparison of manikin versus porcine models in cricothyrotomy procedure training. Emerg Med J. 2008 Nov;25(11):732-4. doi: 10.1136/emj.2008.059014. PMID 18955605
- [Background] Warren JN, Luctkar-Flude M, Godfrey C, Lukewich J. A systematic review of the effectiveness of simulation-based education on satisfaction and learning outcomes in nurse practitioner programs. Nurse Educ Today. 2016 Nov;46:99-108. doi: 10.1016/j.nedt.2016.08.023. Epub 2016 Aug 25. PMID 27621199
- [Background] Jabaay MJ, Marotta DA, Aita SL, Walker DB, Grcevich LO, Camba V, Nolin JR, Lyons J, Giannini J Jr. Medical Simulation-Based Learning Outcomes in Pre-Clinical Medical Education. Cureus. 2020 Dec 3;12(12):e11875. doi: 10.7759/cureus.11875. PMID 33415028
- [Background] Chan CH, Chan TN, Yuen MC, Tung WK. Evaluation of a simulation-based workshop on clinical performance for emergency physicians and nurses. World J Emerg Med. 2015;6(1):16-22. doi: 10.5847/wjem.j.1920-8642.2015.01.003. PMID 25802561
- [Background] Morton S, Avery P, Kua J, O'Meara M. Success rate of prehospital emergency front-of-neck access (FONA): a systematic review and meta-analysis. Br J Anaesth. 2023 May;130(5):636-644. doi: 10.1016/j.bja.2023.01.022. Epub 2023 Feb 28. PMID 36858888
- [Background] Zink N, Merelman A, Fisher AD, Lauria MJ. Emergency Reflex Action Drills and the Problem with Stress. J Spec Oper Med. 2023 Mar 15;23(1):54-58. doi: 10.55460/RCF2-CXS9. PMID 36764288
- [Background] Smith JE, Rickard A, Wise D. Traumatic cardiac arrest. J R Soc Med. 2015 Jan;108(1):11-6. doi: 10.1177/0141076814560837. PMID 25572990
- [Background] Burns KJ, Robinson K, Lowe EG. Evaluation of responses of an air medical helicopter program during a comprehensive emergency response drill. Air Med J. 2007 May-Jun;26(3):139-43. doi: 10.1016/j.amj.2006.08.009. PMID 17467567
- [Background] Anderson NE, Gott M, Slark J. Beyond prognostication: ambulance personnel's lived experiences of cardiac arrest decision-making. Emerg Med J. 2018 Apr;35(4):208-213. doi: 10.1136/emermed-2017-206743. Epub 2018 Jan 5. PMID 29305380
- [Background] Chrimes N. The Vortex: a universal 'high-acuity implementation tool' for emergency airway management. Br J Anaesth. 2016 Sep;117 Suppl 1:i20-i27. doi: 10.1093/bja/aew175. Epub 2016 Jul 20. PMID 27440673
- [Background] Reardon RF, Robinson AE, Kornas R, Ho JD, Anzalone B, Carlson J, Levy M, Driver B. Prehospital Surgical Airway Management: An NAEMSP Position Statement and Resource Document. Prehosp Emerg Care. 2022;26(sup1):96-101. doi: 10.1080/10903127.2021.1995552. PMID 35001821
- [Background] Wang HE, Mann NC, Mears G, Jacobson K, Yealy DM. Out-of-hospital airway management in the United States. Resuscitation. 2011 Apr;82(4):378-85. doi: 10.1016/j.resuscitation.2010.12.014. Epub 2011 Feb 1. PMID 21288624
- [Background] Schauer SG, Naylor JF, Maddry JK, Beaumont DM, Cunningham CW, Blackburn MB, April MD. Prehospital Airway Management in Iraq and Afghanistan: A Descriptive Analysis. South Med J. 2018 Dec;111(12):707-713. doi: 10.14423/SMJ.0000000000000906. PMID 30512120
- [Background] Mabry RL, Frankfurt A. An analysis of battlefield cricothyrotomy in Iraq and Afghanistan. J Spec Oper Med. 2012 Spring;12(1):17-23. doi: 10.55460/FYQG-8E49. PMID 22427045
- [Background] Mabry RL, Edens JW, Pearse L, Kelly JF, Harke H. Fatal airway injuries during Operation Enduring Freedom and Operation Iraqi Freedom. Prehosp Emerg Care. 2010 Apr-Jun;14(2):272-7. doi: 10.3109/10903120903537205. PMID 20199236
- [Background] Brown CA 3rd, Cox K, Hurwitz S, Walls RM. 4,871 Emergency airway encounters by air medical providers: a report of the air transport emergency airway management (NEAR VI: "A-TEAM") project. West J Emerg Med. 2014 Mar;15(2):188-93. doi: 10.5811/westjem.2013.11.18549. PMID 24672610
- See also: Link to information about Student Satisfaction and Self-confidence in Learning, Educational Practices Questionnaire and Simulation Design Scale — https://www.nln.org/education/teaching-resources/tools-and-instruments